CLINICAL TRIAL: NCT04372979
Title: Evaluation Of Efficacy Of COVID-19 Convalescent Plasma Versus Standard Plasma In The Early Care Of COVID-19 Patients Hospitalized Outside Intensive Care Units.
Brief Title: Efficacy of Convalescent Plasma Therapy in the Early Care of COVID-19 Patients.
Acronym: PLASCOSSA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Reluctance of patients and physicians in this transfusion study setting. Blood products have expired. New variants have appeared since the plasma collection period. Some recent publications question the effectiveness of transfusion.
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-A01166-33
Record Dates: First submitted 2020-04-24; First posted 2020-05-04 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; COVID 19; Convalescent plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SARS-CoV-2 patients treated with convalescent plasma (Experimental): Subjects will receive an intravenous injection of SARS-CoV-2 Convalescent Plasma.
  Interventions: Drug: Transfusion of SARS-CoV-2 Convalescent Plasma.
- SARS-CoV-2 patients treated with standard plasma (Active Comparator): Subjects will receive an intravenous injection of standard Plasma.
  Interventions: Drug: Transfusion of standard Plasma.

INTERVENTIONS:
Drug: Transfusion of SARS-CoV-2 Convalescent Plasma. — 2 Convalescent Plasma units of 200-230mL each, inactivated by amotosalen.
  Arms: SARS-CoV-2 patients treated with convalescent plasma
Drug: Transfusion of standard Plasma. — 2 Standard Plasma units of 200-230mL each, inactivated by amotosalen.
  Arms: SARS-CoV-2 patients treated with standard plasma

SUMMARY:
COVID-19 (Corona Virus Disease 2019) hospitalized patients evolution is marked by the risk of worsening of the respiratory system during the second week of the disease. To date, treatments are currently being evaluated and none of them have shown to be effective in the care of these patients. The use of convalescent plasma is a passive immunotherapy. It has often been used in respiratory virus epidemic situations (during the 1918 or 2009 influenza pandemic, or during SARS-CoV-1 or MERS-CoV pandemic). Effects reported in literature are in favour of a beneficial impact of transfusion of these plasma without serious adverse effects reported.

PlasCoSSA is a randomized, controlled, triple-blinded, parallel clinical trial. This study tests the efficacy of convalescent plasma transfusion therapy in the early care of COVID-19 hospitalized patients outside intensive care units.

DETAILED DESCRIPTION:
During SARS-CoV-2 infection, two clinical-biological phases can be observed: an initial viral phase followed by an immunological phase whose onset has been associated with more severe prognosis. Hospitalized patients with comorbidities or clinical risk factors have a higher risk of respiratory functions deterioration and significant risk to need intensive care.

Early transfusion of convalescent plasma (2 units of 200-230 mL of apheresis plasma inactivated by amotosalen) would prevent this secondary worsening and reduce the risk to be transferred to intensive care, length of stay and mortality. Considering clinical and biological manifestations of the disease, including coagulation disorders, endothelial alterations, immunological disorders, it seems interesting to compare this convalescent plasma with a SARS-CoV-2 lacking antibodies plasma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-90 years ;
2. COVID-19 confirmed case ;
3. Cases showing respiratory symptoms, checking at least one of the following criteria:

   1. Cough, dyspnea, respiratory rate > 24 breaths/min
   2. Oxygen saturation < 95% at rest in ambient air
   3. PaO2 < 70mmHg
   4. Scanographic pulmonary compatible with COVID in the absence of any other etiology
4. Risk of deterioration, checking at least one of the following comorbidity criteria :

   1. Chronic respiratory pathology
   2. Diabetes
   3. Cancer pathology
   4. Cardiovascular disease
   5. Chronic kidney failure
   6. Congenital or acquired immunodeficiency
   7. Cirrhosis at stage B
   8. Major sickle cell syndrome
   9. BMI > 30 kg/m2

OR one of the biological criteria :

1. D-dimer 1 µg/mL,
2. Lymphocytes < 0.8 G/L,
3. Ferritin > 300 µg/L,
4. Troponin I > 11 pg/mL or Troponin T > 24.8 pg/mL

Exclusion Criteria:

* Patients admitted in intensive care within the first 6 hours of hospital care,
* Patients after 10 days from the start of symptoms
* Age < 18 years and > 90 years
* Long-term oxygen-dependent patients (at home),
* Decompensated chronic cardiac, respiratory, urological pathology
* Patient refusing administration of blood products,
* Allergic reaction to plasma products,
* IgA deficiency,
* Contraindication to transfusion
* Ig transfusion within 30 days,
* Patient currently participating to another clinical trial,
* Pregnant women,
* No affiliated to the social security,
* Person deprived of liberty by a legal or administrative decision, person under guardianship

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Survival time without needs of a ventilator. | Day 30
  Survival time without needs of ventilator, i.e. the time until oxygen supply (patient previously in ambient air), or an increase by more than 6L/min of O2 for more than 24 hours, or the use of non-invasive ventilation, or intubation, or death.

SECONDARY OUTCOMES:
Morbidity | Day 15
  The percentage of patients i) not hospitalized, without limitation of activities, ii) Not hospitalized, with activity limitation, iii) Hospitalized without oxygen therapy, iv) Hospitalized with oxygen therapy, v) Hospitalized with intensive oxygen therapy or non- invasive ventilation (NIV), vi) Hospitalized and intubated or on extracorporeal membrane oxygenation (ECMO), vii) Dead.
Morbidity | Day 30
  Difference of the SOFA (Sequential Organ Failure Assessment) mean score per patient between the two groups.
Mortality | Day 30
Length of stay | Day 30
Effect on viral pharyngeal specimen clearance | At inclusion and Day 7
  Quantitative SARS-CoV2 PCR carried out on pharyngeal specimen.
Effect on viral blood specimen clearance | At inclusion and Day 7
  Quantitative SARS-CoV2 PCR carried out on blood specimen.
Effect on hemostasis disorders | At inclusion, Day 1 and every 48 hours
  Effects on biological hemostasis parameters disorders.
Kinetics of appearance of neutralizing antibodies | At inclusion, Day 7
  Anti-SARS-Cov2 immunoglobulin G/A level and anti-SARS-Cov2 neutralizing antibody levels.
Transfusion endotheliopathy effect | At inclusion, Day 1, Day 7
  Evolution of biological endotheliopathy parameters
Transfusion biological Inflammation effect | At inclusion, Day 1, Day 7
  Evaluation of biological dosages on inflammation effects
Transfusion hemovigilance | 30 days
  Number of transfusion adverse events
Decrease in the consumption of antibiotics | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie KOULMANN, Study Director — Direction Centrale du Service de Santé des Armées (DCSSA); Catherine VERRET, Study Director — Service de Santé des Armées-Direction de la Formation de la Recherche et de l'Innovation; Christophe MARTINAUD, Principal Investigator — Centre de Transfusion Sanguine des Armées; Jean-Luc BOSSON, Principal Investigator — Statistical and methodological investigator - Laboratoire TIMC UMR 5525 CNRS Equipe Themas
Locations (4):
- France (4):
  - HIA Percy, Clamart
  - HIA Laveran, Marseille
  - HIA Bégin, Saint-Mandé
  - HIA Sainte Anne, Toulon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Ahn DG, Shin HJ, Kim MH, Lee S, Kim HS, Myoung J, Kim BT, Kim SJ. Current Status of Epidemiology, Diagnosis, Therapeutics, and Vaccines for Novel Coronavirus Disease 2019 (COVID-19). J Microbiol Biotechnol. 2020 Mar 28;30(3):313-324. doi: 10.4014/jmb.2003.03011. PMID 32238757
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Zhang B, Liu S, Tan T, Huang W, Dong Y, Chen L, Chen Q, Zhang L, Zhong Q, Zhang X, Zou Y, Zhang S. Treatment With Convalescent Plasma for Critically Ill Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Infection. Chest. 2020 Jul;158(1):e9-e13. doi: 10.1016/j.chest.2020.03.039. Epub 2020 Mar 31. PMID 32243945
- [Background] Walls AC, Park YJ, Tortorici MA, Wall A, McGuire AT, Veesler D. Structure, Function, and Antigenicity of the SARS-CoV-2 Spike Glycoprotein. Cell. 2020 Apr 16;181(2):281-292.e6. doi: 10.1016/j.cell.2020.02.058. Epub 2020 Mar 9. PMID 32155444
- [Background] Zhang JS, Chen JT, Liu YX, Zhang ZS, Gao H, Liu Y, Wang X, Ning Y, Liu YF, Gao Q, Xu JG, Qin C, Dong XP, Yin WD. A serological survey on neutralizing antibody titer of SARS convalescent sera. J Med Virol. 2005 Oct;77(2):147-50. doi: 10.1002/jmv.20431. PMID 16121363
- [Background] Subbarao K, McAuliffe J, Vogel L, Fahle G, Fischer S, Tatti K, Packard M, Shieh WJ, Zaki S, Murphy B. Prior infection and passive transfer of neutralizing antibody prevent replication of severe acute respiratory syndrome coronavirus in the respiratory tract of mice. J Virol. 2004 Apr;78(7):3572-7. doi: 10.1128/jvi.78.7.3572-3577.2004. PMID 15016880
- [Background] Ko JH, Seok H, Cho SY, Ha YE, Baek JY, Kim SH, Kim YJ, Park JK, Chung CR, Kang ES, Cho D, Muller MA, Drosten C, Kang CI, Chung DR, Song JH, Peck KR. Challenges of convalescent plasma infusion therapy in Middle East respiratory coronavirus infection: a single centre experience. Antivir Ther. 2018;23(7):617-622. doi: 10.3851/IMP3243. Epub 2018 Jun 20. PMID 29923831
- [Background] Guo L, Ren L, Yang S, Xiao M, Chang D, Yang F, Dela Cruz CS, Wang Y, Wu C, Xiao Y, Zhang L, Han L, Dang S, Xu Y, Yang QW, Xu SY, Zhu HD, Xu YC, Jin Q, Sharma L, Wang L, Wang J. Profiling Early Humoral Response to Diagnose Novel Coronavirus Disease (COVID-19). Clin Infect Dis. 2020 Jul 28;71(15):778-785. doi: 10.1093/cid/ciaa310. PMID 32198501
- [Background] Thevarajan I, Nguyen THO, Koutsakos M, Druce J, Caly L, van de Sandt CE, Jia X, Nicholson S, Catton M, Cowie B, Tong SYC, Lewin SR, Kedzierska K. Breadth of concomitant immune responses prior to patient recovery: a case report of non-severe COVID-19. Nat Med. 2020 Apr;26(4):453-455. doi: 10.1038/s41591-020-0819-2. No abstract available. PMID 32284614
- [Background] Bouadma L, Lescure FX, Lucet JC, Yazdanpanah Y, Timsit JF. Severe SARS-CoV-2 infections: practical considerations and management strategy for intensivists. Intensive Care Med. 2020 Apr;46(4):579-582. doi: 10.1007/s00134-020-05967-x. Epub 2020 Feb 26. No abstract available. PMID 32103284
- [Background] To KK, Tsang OT, Leung WS, Tam AR, Wu TC, Lung DC, Yip CC, Cai JP, Chan JM, Chik TS, Lau DP, Choi CY, Chen LL, Chan WM, Chan KH, Ip JD, Ng AC, Poon RW, Luo CT, Cheng VC, Chan JF, Hung IF, Chen Z, Chen H, Yuen KY. Temporal profiles of viral load in posterior oropharyngeal saliva samples and serum antibody responses during infection by SARS-CoV-2: an observational cohort study. Lancet Infect Dis. 2020 May;20(5):565-574. doi: 10.1016/S1473-3099(20)30196-1. Epub 2020 Mar 23. PMID 32213337
- [Background] Liu L, Wei Q, Lin Q, Fang J, Wang H, Kwok H, Tang H, Nishiura K, Peng J, Tan Z, Wu T, Cheung KW, Chan KH, Alvarez X, Qin C, Lackner A, Perlman S, Yuen KY, Chen Z. Anti-spike IgG causes severe acute lung injury by skewing macrophage responses during acute SARS-CoV infection. JCI Insight. 2019 Feb 21;4(4):e123158. doi: 10.1172/jci.insight.123158. eCollection 2019 Feb 21. PMID 30830861
- [Background] Tirado SM, Yoon KJ. Antibody-dependent enhancement of virus infection and disease. Viral Immunol. 2003;16(1):69-86. doi: 10.1089/088282403763635465. PMID 12725690
- [Background] Chaichana P, Okabayashi T, Puiprom O, Sasayama M, Sasaki T, Yamashita A, Ramasoota P, Kurosu T, Ikuta K. Low levels of antibody-dependent enhancement in vitro using viruses and plasma from dengue patients. PLoS One. 2014 Mar 18;9(3):e92173. doi: 10.1371/journal.pone.0092173. eCollection 2014. PMID 24642752
- [Background] Houser KV, Broadbent AJ, Gretebeck L, Vogel L, Lamirande EW, Sutton T, Bock KW, Minai M, Orandle M, Moore IN, Subbarao K. Enhanced inflammation in New Zealand white rabbits when MERS-CoV reinfection occurs in the absence of neutralizing antibody. PLoS Pathog. 2017 Aug 17;13(8):e1006565. doi: 10.1371/journal.ppat.1006565. eCollection 2017 Aug. PMID 28817732
- [Background] van Griensven J, Edwards T, de Lamballerie X, Semple MG, Gallian P, Baize S, Horby PW, Raoul H, Magassouba N, Antierens A, Lomas C, Faye O, Sall AA, Fransen K, Buyze J, Ravinetto R, Tiberghien P, Claeys Y, De Crop M, Lynen L, Bah EI, Smith PG, Delamou A, De Weggheleire A, Haba N; Ebola-Tx Consortium. Evaluation of Convalescent Plasma for Ebola Virus Disease in Guinea. N Engl J Med. 2016 Jan 7;374(1):33-42. doi: 10.1056/NEJMoa1511812. PMID 26735992
- [Background] Dufour-Gaume F, Delaune D, Martinaud C, Sailliol A. Early and repeated use of plasma for the management of Ebola patients: Reflection around a case. Transfus Clin Biol. 2017 Feb;24(1):5-8. doi: 10.1016/j.tracli.2016.08.005. Epub 2016 Sep 14. PMID 27640108
- [Background] Tirumalai RS, Chan KC, Prieto DA, Issaq HJ, Conrads TP, Veenstra TD. Characterization of the low molecular weight human serum proteome. Mol Cell Proteomics. 2003 Oct;2(10):1096-103. doi: 10.1074/mcp.M300031-MCP200. Epub 2003 Aug 13. PMID 12917320
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Lippi G, Plebani M. Laboratory abnormalities in patients with COVID-2019 infection. Clin Chem Lab Med. 2020 Jun 25;58(7):1131-1134. doi: 10.1515/cclm-2020-0198. No abstract available. PMID 32119647
- [Background] Sperry JL, Guyette FX, Brown JB, Yazer MH, Triulzi DJ, Early-Young BJ, Adams PW, Daley BJ, Miller RS, Harbrecht BG, Claridge JA, Phelan HA, Witham WR, Putnam AT, Duane TM, Alarcon LH, Callaway CW, Zuckerbraun BS, Neal MD, Rosengart MR, Forsythe RM, Billiar TR, Yealy DM, Peitzman AB, Zenati MS; PAMPer Study Group. Prehospital Plasma during Air Medical Transport in Trauma Patients at Risk for Hemorrhagic Shock. N Engl J Med. 2018 Jul 26;379(4):315-326. doi: 10.1056/NEJMoa1802345. PMID 30044935
- [Background] Chen L, Li X, Chen M, Feng Y, Xiong C. The ACE2 expression in human heart indicates new potential mechanism of heart injury among patients infected with SARS-CoV-2. Cardiovasc Res. 2020 May 1;116(6):1097-1100. doi: 10.1093/cvr/cvaa078. Erratum In: Cardiovasc Res. 2020 Oct 1;116(12):1994. doi: 10.1093/cvr/cvaa157. PMID 32227090
- [Background] Recalcati S. Cutaneous manifestations in COVID-19: a first perspective. J Eur Acad Dermatol Venereol. 2020 May;34(5):e212-e213. doi: 10.1111/jdv.16387. No abstract available. PMID 32215952
- [Background] Wu F, Peng Z, Park PW, Kozar RA. Loss of Syndecan-1 Abrogates the Pulmonary Protective Phenotype Induced by Plasma After Hemorrhagic Shock. Shock. 2017 Sep;48(3):340-345. doi: 10.1097/SHK.0000000000000832. PMID 28107214
- [Background] Whitney JE, Zhang B, Koterba N, Chen F, Bush J, Graham K, Lacey SF, Melenhorst JJ, Teachey DT, Mensinger JL, Yehya N, Weiss SL. Systemic Endothelial Activation Is Associated With Early Acute Respiratory Distress Syndrome in Children With Extrapulmonary Sepsis. Crit Care Med. 2020 Mar;48(3):344-352. doi: 10.1097/CCM.0000000000004091. PMID 32058372
- [Background] Garraud O, Heshmati F, Pozzetto B, Lefrere F, Girot R, Saillol A, Laperche S. Plasma therapy against infectious pathogens, as of yesterday, today and tomorrow. Transfus Clin Biol. 2016 Feb;23(1):39-44. doi: 10.1016/j.tracli.2015.12.003. Epub 2016 Jan 6. PMID 26775794
- [Background] Dinsdale RJ, Hazeldine J, Al Tarrah K, Hampson P, Devi A, Ermogenous C, Bamford AL, Bishop J, Watts S, Kirkman E, Dalle Lucca JJ, Midwinter M, Woolley T, Foster M, Lord JM, Moiemen N, Harrison P. Dysregulation of the actin scavenging system and inhibition of DNase activity following severe thermal injury. Br J Surg. 2020 Mar;107(4):391-401. doi: 10.1002/bjs.11310. Epub 2019 Sep 10. PMID 31502663
- [Background] Squizzato A, Hunt BJ, Kinasewitz GT, Wada H, Ten Cate H, Thachil J, Levi M, Vicente V, D'Angelo A, Di Nisio M. Supportive management strategies for disseminated intravascular coagulation. An international consensus. Thromb Haemost. 2016 May 2;115(5):896-904. doi: 10.1160/TH15-09-0740. Epub 2015 Dec 17. PMID 26676927
- [Background] Di Nisio M, Thachil J, Squizzato A. Management of disseminated intravascular coagulation: a survey of the International Society on Thrombosis and Haemostasis. Thromb Res. 2015 Aug;136(2):239-42. doi: 10.1016/j.thromres.2015.05.022. Epub 2015 May 23. PMID 26033399
- [Background] Garraud O, Malot S, Herbrecht R, Ojeda-Uribe M, Lin JS, Veyradier A, Payrat JM, Liu K, Corash L, Coppo P. Amotosalen-inactivated fresh frozen plasma is comparable to solvent-detergent inactivated plasma to treat thrombotic thrombocytopenic purpura. Transfus Apher Sci. 2019 Dec;58(6):102665. doi: 10.1016/j.transci.2019.10.007. Epub 2019 Nov 5. PMID 31740165
- [Background] van Griensven J, De Weiggheleire A, Delamou A, Smith PG, Edwards T, Vandekerckhove P, Bah EI, Colebunders R, Herve I, Lazaygues C, Haba N, Lynen L. The Use of Ebola Convalescent Plasma to Treat Ebola Virus Disease in Resource-Constrained Settings: A Perspective From the Field. Clin Infect Dis. 2016 Jan 1;62(1):69-74. doi: 10.1093/cid/civ680. Epub 2015 Aug 10. PMID 26261205
- [Background] Brown JF, Dye JM, Tozay S, Jeh-Mulbah G, Wohl DA, Fischer WA 2nd, Cunningham CK, Rowe K, Zacharias P, van Hasselt J, Norwood DA, Thielman NM, Zak SE, Hoover DL. Anti-Ebola Virus Antibody Levels in Convalescent Plasma and Viral Load After Plasma Infusion in Patients With Ebola Virus Disease. J Infect Dis. 2018 Jul 13;218(4):555-562. doi: 10.1093/infdis/jiy199. PMID 29659889
- [Background] Di Minno G, Navarro D, Perno CF, Canaro M, Gurtler L, Ironside JW, Eichler H, Tiede A. Pathogen reduction/inactivation of products for the treatment of bleeding disorders: what are the processes and what should we say to patients? Ann Hematol. 2017 Aug;96(8):1253-1270. doi: 10.1007/s00277-017-3028-4. Epub 2017 Jun 18. PMID 28624906
- [Background] Ahn JY, Sohn Y, Lee SH, Cho Y, Hyun JH, Baek YJ, Jeong SJ, Kim JH, Ku NS, Yeom JS, Roh J, Ahn MY, Chin BS, Kim YS, Lee H, Yong D, Kim HO, Kim S, Choi JY. Use of Convalescent Plasma Therapy in Two COVID-19 Patients with Acute Respiratory Distress Syndrome in Korea. J Korean Med Sci. 2020 Apr 13;35(14):e149. doi: 10.3346/jkms.2020.35.e149. PMID 32281317
- [Background] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Soo YO, Cheng Y, Wong R, Hui DS, Lee CK, Tsang KK, Ng MH, Chan P, Cheng G, Sung JJ. Retrospective comparison of convalescent plasma with continuing high-dose methylprednisolone treatment in SARS patients. Clin Microbiol Infect. 2004 Jul;10(7):676-8. doi: 10.1111/j.1469-0691.2004.00956.x. PMID 15214887
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Shi Y, Wang Y, Shao C, Huang J, Gan J, Huang X, Bucci E, Piacentini M, Ippolito G, Melino G. COVID-19 infection: the perspectives on immune responses. Cell Death Differ. 2020 May;27(5):1451-1454. doi: 10.1038/s41418-020-0530-3. Epub 2020 Mar 23. No abstract available. PMID 32205856
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Chang L, Yan Y, Wang L. Coronavirus Disease 2019: Coronaviruses and Blood Safety. Transfus Med Rev. 2020 Apr;34(2):75-80. doi: 10.1016/j.tmrv.2020.02.003. Epub 2020 Feb 21. PMID 32107119
- [Background] Hashem AM, Hassan AM, Tolah AM, Alsaadi MA, Abunada Q, Damanhouri GA, El-Kafrawy SA, Picard-Maureau M, Azhar EI, Hindawi SI. Amotosalen and ultraviolet A light efficiently inactivate MERS-coronavirus in human platelet concentrates. Transfus Med. 2019 Dec;29(6):434-441. doi: 10.1111/tme.12638. Epub 2019 Nov 6. PMID 31696565
- [Background] Lin L, Hanson CV, Alter HJ, Jauvin V, Bernard KA, Murthy KK, Metzel P, Corash L. Inactivation of viruses in platelet concentrates by photochemical treatment with amotosalen and long-wavelength ultraviolet light. Transfusion. 2005 Apr;45(4):580-90. doi: 10.1111/j.0041-1132.2005.04316.x. PMID 15819680
- [Background] Chang L, Zhao L, Gong H, Wang L, Wang L. Severe Acute Respiratory Syndrome Coronavirus 2 RNA Detected in Blood Donations. Emerg Infect Dis. 2020 Jul;26(7):1631-1633. doi: 10.3201/eid2607.200839. Epub 2020 Jun 21. PMID 32243255
- See also: Anticoagulant treatment for the prevention of thrombotic risk in a patient hospitalized with COVID-19 and monitoring of hemostasis. — https://sfar.org/download/traitement-anticoagulant-pour-la-prevention-du-risque-thrombotique-chez-un-patient-hospitalise-avec-covid-19-et-surveillance-de-lhemostase/
- See also: Efficacy and Safety Human Coronavirus Immune Plasma (HCIP) vs. Control (SARS-CoV-2 Non-immune Plasma) Among Adults Exposed to COVID-19 - Full Text View - ClinicalTrials.gov — https://clinicaltrials.gov/ct2/show/NCT04323800
- See also: Transfusion of therapeutic plasma: products, indications (Haute Autorité de Santé, France) — https://www.has-sante.fr/jcms/c_1264081/fr/transfusion-de-plasma-therapeutique-produits-indications
- See also: Coronavirus SARS-CoV-2 management of people at risk of severe forms (Haut Conseil de la Santé Publique; 2020) — https://www.hcsp.fr/explore.cgi/avisrapportsdomaine?clefr=790